CLINICAL TRIAL: NCT04070092
Title: The Impact of Traumatic Brain Injury in the Elderly: a Prospective Study
Brief Title: The Impact of Traumatic Brain Injury in the Elderly
Status: Suspended | Type: Observational
Why Stopped: Search for new funding
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Principal Investigator, prof. dr. Bart Depreitere, clinical professor, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S62845
Record Dates: First submitted 2019-08-23; First posted 2019-08-28 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Traumatic Brain Injury
Keywords: Traumatic Brain Injury; Elderly; Cognitive Impairment; Motor impairment; Brain injury; Quality of life; Impact; Health care economic costs
MeSH Terms: conditions — Brain Injuries, Traumatic; Cognitive Dysfunction; Brain Injuries; Tooth, Impacted

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples Without DNA — Blood samples for biomarkers study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI group: A cohort of patients admitted to UZ Leuven from 2019 to 2023 due to Traumatic Brain Injury and fulfilling our inclusion and exclusion criteria will be recruited.
  * Inclusion criteria will be: ≥ 65 years old, admitted to UZ Leuven between 2019 and 2023 due to TBI, all injury severities (mild (GCS 13-15), moderate (GCS 9-12) or severe (GCS ≤8)), and having signed the informed consent to participate in the study.
  * Exclusion criteria will be: < 65 years old, admitted to UZ Leuven before 2019, diagnose of neurodegenerative diseases before the TBI, cognitive and motor disturbances caused by any other pathology, previous alcohol/drugs abuse, and not having signed the informed consent to participate in the study.
- Control group: A cohort of healthy volunteers with similar demographic characteristics will be recruited as a control group.
  * Inclusion criteria will be: ≥ 65 years old and having signed the informed consent to participate in the study.
  * Exclusion criteria will be: < 65 years old, diagnose of neurodegenerative diseases, cognitive and motor disturbances caused by any pathology, previous alcohol/drugs abuse, and not having signed the informed consent to participate in the study.

SUMMARY:
A better understanding of the impact of Traumatic Brain Injury (TBI) in the elderly, in terms of brain damage, cognitive and motor functions, sleep quality and quality of life is necessary due to the increasing incidence and prevalence of TBI in this population and its high economic impact on society. Therefore, this study aims at describing the short-term consequences of TBI by studying injury patterns, injury severity, risk profiles, brain damage, co-morbidities, post-traumatic history, level of dependency, serum-based injury biomarkers, cognitive and motor functions, sleep quality and quality of life 6 months after TBI. All the obtained results will be integrated in a new prognostic tool for the course of the outcomes of TBI in the elderly population.

DETAILED DESCRIPTION:
In order to achieve the goals of the project, a cohort of 50 patients and 50 volunteers is expected, and the following evaluations will be performed:

For the patients group, after signing the informed consent form, a clinical data collection, a serum-based injury biomarkers study, a brain damage assessment, a cognitive and motor assessment, a sleep quality and a quality of life evaluation will be performed.

* Data collection: injury patterns, injury severity, co-morbidities and post-traumatic history will be prospectively registered in our cohort of patients in order to study which types of accidents are risky to result in poor outcome. This will be done through the data collection in medical records of the patients. Advanced statistical methods, such as Gaussian models, will be applied in order to find relations between input and outcome to the best extent possible. In addition, injury mechanisms will be categorized into classes with more or less similar magnitudes of force and acceleration inputs.
* Serum based injury biomarkers study: blood samples from our cohort, taken by UZ Leuven nurses in the context of routine-clinical practice will be studied by the Laboratory for Molecular Neurobiomarker Research in UZ Leuven, through Enzyme-Linked Immunosorbent Assay (ELISA). No data will be available for the control group. The results will be compared to results previously obtained in the Laboratory for Molecular Neurobiomarker Research from healthy patients with similar demographic characteristics.
* CT imaging: CT images performed in the context of routine clinical practice at admission and follow up will be obtained from the hospital's database. The scans will be carefully studied, using automated reports created by Icometrix and the Marshall Head Injury Scale, in order to quantify brain damage. No data will be available for the control group, so results will not be compared between both groups. These findings will be related with the results obtained in the serum-based injury biomarkers study and cognitive and motor assessments.
* Economic impact prospective analysis: hospital costs for the clinical management in our cohort will be extracted from the financial database of UZ Leuven, in order to know what is the economic impact that TBI in the elderly has on society.

  1st evaluation session with the patient: 6 months after the injury, the patient will be called back to UZ Leuven for evaluation.The protocol for this session will be done in 1 or 2 sessions, depending on the preferences of the patient, and will consist of:
* MRI: High-resolution T1 and T2 weighted imaging sequences will be used to study volumetric and morphological changes in the brain. Moreover, Diffusion Tractography Imaging (DTI) will be used to study changes in white matter. Susceptibility Weighted Imaging (SWI) sequences will also be included in order to study axonal injuries and microbleeds. One MRI scan will be obtained from each patient and the results will be interpreted with the Icobrain TBI report, provided by Icometrix.
* Cognitive assessment: the CANTAB test will be used to study cognitive functions after TBI, as it is a validated and reliable computerized neuropsychological battery, consisting of memory, learning, attention, problem solving and executive function test. Moreover, the patients' level of education will be asked, registered and correlated with the results obtained in our evaluations.
* Motor assessment: it will be performed using the Berg Balance Scale (BBS), Timed Up an Go (TUG) test, Timed Up and Go with cognitive dual task (TUGcog) test, Box-and-block test and a cycling test performed with a bicycle simulator created by the IMPAct group (KU Leuven).
* Sleep quality assessment: the sleep quality in our cohort will be assessed using the Pittsburgh Sleep Quality Index, in order to understand how TBI can affect the patients' sleep patterns.
* Quality of life evaluation: the quality of life in our cohort will be assessed with the Quality of Life after Brain Injury (QOLIBRI) tool, in the same session as cognitive and motor outcomes, in order to understand how the quality of life is affected in the elderly population after TBI.

All the results will be compared with the results obtained in the control group.

If the patient chooses to have two evaluation sessions, instead of one, the first session will be dedicated to the MRI scan and the second session will be dedicated to the cognitive, motor, sleep quality and quality of life evaluation. Both sessions will be performed within the same week.

For the control group, after signing the informed consent form MRI scans, a cognitive and motor assessment, sleep quality and quality of life evaluation will be performed in this group at the time of recruitment, in one or two sessions, depending on the preference of the volunteer. All the assessments will be performed in University Hospitals Leuven and the results will be compared with the patients group's results.

* MRI: High-resolution T1 and T2 weighted imaging sequences will be used to study volumetric and morphological changes in the brain. Moreover, Diffusion Tractography Imaging (DTI) will be used to study changes in white matter. Susceptibility Weighted Imaging (SWI) sequences will also be included in order to study axonal injuries and microbleeds . One MRI scan will be obtained from each volunteer and the results will be interpreted with the Icobrain TBI report, provided by Icometrix, and compared with the results obtained for the patients.
* Cognitive assessment: CANTAB test will be used to study cognitive functions in this group, as it is a validated and reliable computerized neuropsychological battery, consisting of memory, learning, attention, problem solving and executive function test. Moreover, the volunteers level of education will be asked, registered and correlated with the results obtained in our evaluations.
* Motor assessment: it will be performed using the Berg Balance Scale (BBS), Timed Up an Go (TUG) test, Timed Up and Go with cognitive dual task (TUGcog) test, Box-and-block test and a cycling test performed with a bicycle simulator created by the IMPAct group (KU Leuven).
* Sleep quality assessment: the sleep quality in our cohort will be assessed using the Pittsburgh Sleep Quality Index.
* Quality of life evaluation: the quality of life in this group will be assessed with the Quality of Life after Brain Injury (QOLIBRI) tool, in the same session as cognitive and motor outcomes, in order to understand how the quality of life is affected in the elderly population after TBI.

If the volunteer chooses to have two evaluation sessions, instead of one, the first session will be dedicated to the MRI scan and the second session will be dedicated to the cognitive, motor, sleep quality and quality of life evaluation. Both sessions will be performed within the same week.

ELIGIBILITY:
Inclusion Criteria for patients:

* ≥ 65 years old
* admitted to UZ Leuven between 2019 and 2023 due to TBI
* all injury severities (mild (GCS 13-15), moderate (GCS 9-12) or severe (GCS ≤8))
* having signed the informed consent to participate in the study.

Inclusion Criteria for healthy volunteers:

* ≥ 65 years old
* having signed the informed consent to participate in the study.

Exclusion Criteria for patients:

* < 65 years old, admitted to UZ Leuven before 2019
* diagnose of neurodegenerative diseases before the TBI
* cognitive and motor disturbances caused by any other pathology
* previous alcohol/drugs abuse
* not having signed the informed consent to participate in the study.

Exclusion criteria for the healthy volunteers will be:

* < 65 years old
* diagnose of neurodegenerative diseases
* cognitive and motor disturbances caused by any pathology
* previous alcohol/drugs abuse
* not having signed the informed consent to participate in the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: A cohort of patients ≥65 years old admitted to UZ Leuven between 2019 and 2023 due to TBI (patients group) and a cohort of healthy volunteers with similar demographic characteristics (control group) will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Data collection | September 2019-December 2022
  Injury patterns, injury severity, co-morbidities and post-traumatic history will be prospectively registered in our cohort of patients in order to study which types of accidents are risky to result in poor outcome. This will be done through the data collection in medical records of the patients. Advanced statistical methods, such as Gaussian models, will be applied in order to find relations between input and outcome to the best extent possible. In addition, injury mechanisms will be categorized into classes with more or less similar magnitudes of force and acceleration inputs.
Serum based injury biomarkers study | September 2019-December 2022
  Blood samples from our cohort, taken by UZ Leuven nurses in the context of routine-clinical practice will be studied by the Laboratory for Molecular Neurobiomarker Research in UZ Leuven, through Enzyme-Linked Immunosorbent Assay (ELISA). No data will be available for the control group. The results will be compared to results previously obtained in the Laboratory for Molecular Neurobiomarker Research from healthy patients with similar demographic characteristics.
CT imaging | September 2019-December 2022
  CT images performed in the context of routine clinical practice at admission and follow up will be obtained from the hospital's database. The scans will be carefully studied, using automated reports created by Icometrix and the Marshall Head Injury Scale, in order to quantify brain damage. No data will be available for the control group, so results will not be compared between both groups. These findings will be related with the results obtained in the serum-based injury biomarkers study and cognitive and motor assessments.
Economic impact prospective analysis | September 2019-December 2022
  Hospital costs for the clinical management in our cohort will be extracted from the financial database of UZ Leuven, in order to know what is the economic impact that TBI in the elderly has on society.
MRI | September 2019-December 2022
  High-resolution T1 and T2 weighted imaging sequences will be used to study volumetric and morphological changes in the brain. Moreover, Diffusion Tractography Imaging (DTI) will be used to study changes in white matter. Susceptibility Weighted Imaging (SWI) sequences will also be included in order to study axonal injuries and microbleeds. One MRI scan will be obtained from each patient and healthy volunteer.
Cognitive assessment | September 2019-December 2022
  The CANTAB test will be used to study cognitive functions after TBI, as it is a validated and reliable computerized neuropsychological battery, consisting of memory, learning, attention, problem solving and executive function test. Moreover, the patients' level of education will be asked, registered and correlated with the results obtained in our evaluations.
Motor assessment | September 2019-December 2022
  The following motor assessment tests will be used: Berg Balance Scale (BBS), Timed Up an Go (TUG),Timed Up and Go with cognitive dual task (TUGcog), Box-and-block, and a Cycling test with a bicycle simulator created by the IMPAct group (KU Leuven), which evaluate cycling skills.
Quality of life evaluation | September 2019-December 2022
  The quality of life in our cohort will be assessed with the Quality of Life after Brain Injury (QOLIBRI) tool, in the same session as cognitive and motor outcomes, in order to understand how the quality of life is affected in the elderly population after TBI.
Sleep quality assessment | May 2021-December 2022
  The sleep quality in our cohort will be assessed using the Pittsburgh Sleep Quality Index

CONTACTS AND LOCATIONS:
Overall Officials: Bart Depreitere, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No